CLINICAL TRIAL: NCT03214926
Title: A Pilot Study to Evaluate the Augmented Reality-Based Dance Application on Mobility and Balance of Persons With Parkinson's Disease
Brief Title: Moving Through Glass: An Augmented Reality Device Application for Persons With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Syracuse University (Other)
Responsible Party: Principal Investigator, Luis Columna, Associate Professor, Syracuse University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 16239
Record Dates: First submitted 2017-07-07; First posted 2017-07-12 (Actual); Last update posted 2018-12-04 (Actual); Status verified 2018-11

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease; Dance; Google Glass; Mobility; Balance
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Prospective uncontrolled pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Moving Through Glass intervention (Experimental): Participants were asked to use Moving Through Glass (MTG) intervention on Google Glass for at least once a day for 3 weeks. MTG intervention includes 4 difference guided-dance/movement modules for the participants.
  Interventions: Device: Moving Through Glass intervention

INTERVENTIONS:
Device: Moving Through Glass intervention

SUMMARY:
Recently, Mark Morris Dance Group, and created Moving Through Glass (MTG), a project that was funded by Google, as a portable, round-the-clock extension of the internationally acclaimed Dance for Parkinson's Disease (PD)®. When a user activates Glass, participants can choose from a variety of different exercises, like "warm me up" or "balance me." Once selected, they see the founder instructors of the Dance for PD® projected in front of them.

As a single site research study at Syracuse University, researchers are conducting the pilot phase of the research project.

The purpose of the study is to investigate the impact of MTG on quality of life and motor functions (i.e. balance, gait, fall efficacy). Participation in the study required three visits to Women's Building in a period of four weeks and about 1-3 hours of the participant's time at each visit. During the first visit, 1 participants reviewed the consent form, completed Montreal Cognitive Assessment (MOCA) and if qualified participated in a face-to-face interview. Participants were given survey package to fill out at home and were given a week to complete all the paperwork. On the second visit, they returned the completed survey package, were given physical assessments and were taught how to use Google Glass. The participants left with Google Glass, log sheet, and survey package. After 3 weeks, participants came to Women's Building for the last visit and the physical assessments were repeated, followed by an exit interview.

DETAILED DESCRIPTION:
The common symptoms of Parkinson's disease (PD) include but are not limited to resting tremor, muscular rigidity, and difficulty in initiating movement. These motor impairments, which can negatively impact the fluidity and pacing of movement, can increase the risk people with PD face in their daily activities. Additionally, non-motor symptoms such as apathy and depression can often lead to isolation, potentially reducing physical activity in people with PD.

In 2001, Dance for Parkinson's Disease (DfPD), a collaboration between Brooklyn Parkinson Group (BPG) and Mark Morris Dance Group (MMDG), an internationally known company based in Brooklyn, began providing dance classes for the Parkinson community to train other teachers in the hopes of developing cognitive strategies and to enhance the sense of community and the amount of physical activity in PD population. Since then, positive effects of dance in motor and cognitive functions of people with PD have been reported from several types of dance classes.

While recent research has investigated dance as a therapy for people with Parkinson's disease (PD), there is only one study, to our knowledge, that investigates the use of Google Glass as a portable way for persons with PD to use cued movement as they perform activities of daily living to help temporarily alleviate symptoms such as freezing, initiating movement, and balancing. This qualitative study explored the acceptability of the Google Glass in five participants with PD, as well as their caregivers. The results of this study showed that participants highly favored the voice activation system used to control this technology, especially in comparison to the frustrations expressed using touch screen smart phones. The participants also expressed increased confidence because the Google Glass gave them a sense of independence when going out into public alone. Despite the potential beneficial uses of the Glass, due to the highly complicated menus with multiple applications participants found using the Glass frustrating. Additionally, low number of participants used in this study, very short intervention time, and the lack of quantitative data suggests that further investigation of use of a simplified version of Google Glass in rehabilitation of Parkinson's disease is necessary.

Recently, MMDG created Moving Through Glass (MTG), a project that was funded by Google, as a portable, round-the-clock extension of the internationally acclaimed Dance for PD®. When a user activates Glass, they can choose from a variety of different exercises, like "warm me up" or "balance me." Once selected, they see the founder instructors of the Dance for PD® projected in front of them.

As a single site research study at Syracuse University, researchers will be conducting the pilot phase of the research project. MMDG provided the research team with the three pairs of glasses needed to complete this study. At the end of this study, the glasses will be returned to MMDG. The MTG questionnaire (described in detail in Section 4), provided by MMDG as part of their product development, will also be given to the participants to collect information about the product. MTG questionnaires, including only deidentified, gross data, will be shared with MMDG as a part of product development, not research. Researchers will NOT be reporting our research findings to Google or MMDG.

The purpose of the study is to investigate the impact of MTG on quality of life and motor functions (i.e. balance, gait, fall efficacy). Researchers are trying to answer the following questions:

Purpose #1: What are the Parkinson's disease patients' experiences (constraints, benefits, strategies, etc) related to physical activity?

Purpose #2: What is the participants' perception of using Google Glass during their daily activities? In topics related to:

* Perceived competence
* Movement independency
* Participation in physical activity
* Participation in social interactions

Participants in this study will be people with Parkinson's disease. Researchers plan to recruit 15 subjects in this project. Due to the limited number of Google Glasses (3 pairs), only 3 participants will go through the study at a given time period. Once recruited, the participants will be expected to make three visits to Women's Building at Syracuse University in a one-month period. On the first visit, researchers will go over the consent form with the participants. Upon signing the forms, participants will be asked to complete the Montreal Cognitive Assessment (MOCA, 10 min). The MOCA is shown to be a highly sensitive cognitive assessment even for mild cognitive impairment and is used widely with Parkinson's population. Researchers will use this assessment to have a cut-off point for the exclusion criteria for the participants who are in a high-risk group for dementia. The optimal cut-off value of 22 is determined on a 30-point scale, with 30 indicating no cognitive problems. The scale is comprised of 7 sub scores that include executive functioning, memory, naming, attention, language, abstraction, and orientation. If the inclusion criteria are met, the participants will also participate in a face-to-face semi-structured interview to explore their perception regarding movement strategies, fear of falling, patterns of physical recreation, perceived benefits, and constraints. This interview will occur before the implementation of the program. The duration of each interview will be between 60 to 75 minutes. This interview will be audio and video recorded. The purpose of video and audio recording of the interviews is to ensure that we capture the essential meaning of participants' experiences.

Once the interviews are completed, the participants will receive a package that includes several questionnaires and surveys.

ELIGIBILITY:
Inclusion Criteria:

* self-reported diagnosis of Parkinson's disease
* age 18 years or over

Exclusion Criteria:

* Movement Disorder Society-sponsored Unified Parkinson's Disease Rating Scale (MDS-UPDRS) part III> 57
* Montreal Cognitive Assessment (MOCA)<21,
* not being able to wear or operate Google Glass.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-10-17 (Actual); Primary Completion 2017-05-28 (Actual); Study Completion 2017-05-28 (Actual)

PRIMARY OUTCOMES:
Mobility | 3 weeks
  To assess the mobility of people with Parkinson's disease. This outcome will be measured using the Mini Balance Evaluations System Test (Mini-BESTest)

SECONDARY OUTCOMES:
Mood | 3 weeks
  To assess the depression levels of people with Parkinson's disease. This outcome will be measured using the Becks Depression Inventory (BDI)
Quality of life of Participants | 3 weeks
  To assess the quality of life of people with Parkinson's disease. This outcome will be measured using the Parkinson's Disease Quality of Life questionnaire (PDQL)
Google Glass experience-Questionnaire | 3 weeks
  To assess the experiences of persons with PD regarding the Google Glass use. This outcome will be measured using the Moving Through Glass questionnaire.
Quantitative measures of the Google Glass experience | 3 weeks
  To assess the experiences of persons with PD regarding the Google Glass use. This outcome will be measured using quantitative participant report.
Qualitative measures of the Google Glass experience | 3 weeks
  To assess the experiences of persons with PD regarding the Google Glass use. This outcome will be measured using qualitative participant interviews.
Balance-MiniBestTEst | 3 weeks
  To assess the balance of people with Parkinson's disease. This outcome will be measured using the Mini Balance Evaluations System Test (Mini-BESTest)
Balance-ABC | 3 weeks
  To assess the balance of people with Parkinson's disease. This outcome will be measured using the Activity-specific Balance Confidence scale (ABC)
Physical activity | 3 weeks
  To assess the engagement in physical activity of people with Parkinson's disease. This outcome will be measured using the Physical Activity Scale for Elderly (PASE).

CONTACTS AND LOCATIONS:
Overall Officials: Luis Columna, PhD, Principal Investigator — Syracuse University

IPD SHARING:
Plan to Share IPD: No